CLINICAL TRIAL: NCT01930695
Title: Post Market Clinical Follow-up of CRT-DX Therapy With Lumax 640/740 HF-T
Acronym: Pre-CRAFT
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: CR013
Record Dates: First submitted 2013-08-21; First posted 2013-08-29 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: DX functionality; Atrial fibrillation; CRT-D indication
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is designed to collect data of the performance and confirm the safety of the DX (Diagnostic eXtension) functionality in the Lumax 640/470 HF-T in patients with permanent atrial fibrillation and CRT-D indication according to current ESC guidelines. The DX functionality is a feature, which can be activated in the Lumax 640/740 HF-T when connected to the LinoxSMART S DX right ventricular lead. The combination of these devices enable atrial sensing via a sensing dipole in the ventricular lead and therefore reduces the number of implanted leads without sacrificing atrial information. Atrial pacing can not be provided but is not needed in patients with permanent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* CRT-D indication according to current ESC guidelines (NYHA III/IV; QRS≥120ms; LVEF≤35%; Expected survival ≥ 1 year; need for pacing because of slow ventricular rate or pacemaker dependency as a result of AV nodal ablation or ventricular rate ≤60bpm at rest and ≤90bpm on exercise)
* Permanent atrial fibrillation
* Patients planned to be implanted with BIOTRONIK Lumax 640/740 HF-T
* Patients planned to be implanted with BIOTRONIK LinoxSmart S DX right ventricular lead (or successors)
* Patient eligible for programming of DX functionality according to the physicians' decision
* Patient is willing and able to comply with the CIP and provided written informed consent
* Patient accepts Home Monitoring® concept and has sufficient GSM/GPRS coverage

Exclusion Criteria:

* Patients with any contraindication to CRT-D therapy
* Patients listed for heart transplantation
* Life expectancy less than 12 months
* Pregnant or breast-feeding women
* Patients under the age of 18
* Patients with limited contractual capability
* Participation in any other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure patients with CRT-D indication according to current ESC guidelines and permanent atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Quality of IEGM recording | 3 months
  to assess if the IEGM Online recordings of the Lumax 640/740 HF-T with DX functionality provide adequate quality to classify the atrial rhythm
Safety of the Lumax 640/740 HF-T with DX functionality based on the Serious Adverse Device Effects related to the DX functionality | 3 months
  to assess the safety of the Lumax 640/740 HF-T by the analysis of Serious Adverse Device Effects which are related to the DX functionality
Safety of the Lumax 640/740 HF-T with DX functionality based on all, serious and non-serious, Adverse Device Effects related to DX functionality | 3 months
  to assess the safety of the Lumax 640/740 HF-T with DX functionality by the analysis of all (serious and non-serious) Adverse Device Effects which are related to the DX functionality
Number of patients with maintenance of diagnosis of permanent AF | 3 months
  to investigate whether the diagnosis of permanent AF at enrollment is maintained after device implantation

CONTACTS AND LOCATIONS:
Overall Officials: Christian Sticherling, Prof. Dr., Study Chair — Universitätsspital Basel, Petersgraben 4, 4031 Basel, Switzerland
Locations (5):
- Germany (4):
  - Herz- und Gefäßzentrum Bad Bevensen, Bad Bevensen
  - St. Marien-Hospital Lünen, Lünen
  - Deutsches Herzzentrum München, München
  - DRK Mölln-Ratzeburg, Ratzeburg
- Universitätsspital Basel, Basel, Switzerland

REFERENCES:
- [Result] Sticherling C, Muller D, Schaer BA, Kruger S, Kolb C; Pre-CRAFT investigators. Atrial electrogram quality in single-pass defibrillator leads with floating atrial bipole in patients with permanent atrial fibrillation and cardiac resynchronization therapy. Indian Pacing Electrophysiol J. 2018 Jul-Aug;18(4):140-145. doi: 10.1016/j.ipej.2018.03.005. Epub 2018 Mar 27. PMID 29596906